CLINICAL TRIAL: NCT01668680
Title: Metronomic Chemotherapy With Anti-angiogenic Effect as Maintenance Treatment for Metastatic Colorectal Carcinoma Following Response to FOLFIRI+Bevacizumab: Clinical and Laboratory Studies
Brief Title: Maintenance Metronomic Chemotherapy for Metastatic Colorectal Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No satisfactory acrual
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMC-0047-11
Record Dates: First submitted 2012-03-11; First posted 2012-08-20 (Estimated); Last update posted 2015-07-08 (Estimated); Status verified 2015-07

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Metronomic Chemotherapy; Anti-Angiogenic; Maintenance Treatment; Colorectal Cancer Metastatic
MeSH Terms: interventions — Capecitabine; Celecoxib; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LDM anti-angiogenic chemotherapy (Experimental): LDM (Low Dose Metronomic) anti-angiogenic chemotherapy includes daily oral treatment with CAPECITABINE, CELECOXIB and METHOTREXATE.
  Interventions: Drug: CAPECITABINE, CELECOXIB and METHOTREXATE
- observation (No Intervention): observation only

INTERVENTIONS:
Drug: CAPECITABINE, CELECOXIB and METHOTREXATE — daily oral treatment with CAPECITABINE, CELECOXIB and METHOTREXATE
  Other Names: Metronomic Chemotherapy
  Arms: LDM anti-angiogenic chemotherapy

SUMMARY:
Colorectal cancer patients with metastases (mCRC) at response under expensive chemotherapy which may be toxic +/- exhausting are candidates for an effective and more convenient maintenance treatment.

Objectives:

1. To define the efficacy of maintenance chemotherapy by a low-dose metronomic (LDM) regimen, in metastatic CRC patients responding under FOLFIRI + bevacizumab.
2. To discover predictive factors for response to this LDM regimen.

Hypothesis:

1. The re-growth of residual metastases can be slowed by the anti-angiogenic effects of LDM chemotherapy.
2. Serial measurements of angiogenic/ inflammatory factors in the plasma and/or evaluation of certain enzymes in the tumor may discover predictive factors of response to LDM chemotherapy in metastatic CRC patients.

DETAILED DESCRIPTION:
At entry to the research protocol the up-till then administered treatment with Intra Venous FOLFIRI+BEVACIZUMAB will be stopped.Instead, the research oral treatment will be initiated to be taken daily on an ambulatory basis and under once monthly re-evaluation. If and when disease progresses the original FOLFIRI+BEVACIZUMAB treatment will be considered for re-institution.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic (or cytologic) proof of colorectal carcinoma (CRC).
2. Age: between 18 and 80.
3. Sex: both sexes.
4. Previous treatment for metastatic disease is limited to FOLFIRI+ bevacizumab.
5. Prior adjuvant chemotherapy, with a fluoropyrimidine and/or Oxaliplatin, is allowed.
6. Prior radiotherapy, either as adjuvant treatment or palliation of metastatic sites is allowed, provided that there are other non-irradiated foci of disease for evaluation.
7. Persistent remission, either complete, partial or minimal response (CR, PR or MR) or stable disease (SD), one year+/-one month from initiation of first line treatment for mCRC.
8. Asymptomatic patients at break from chemotherapy.
9. Intact organ function, including complete blood counts (CBC) showing normal values or any toxicity limited to grade 1 and blood chemistry (SMA) showing liver and renal functions < 1.5 upper normal limit (UNL).
10. Capability to understand and to sign the informed consent.

Exclusion Criteria:

1. Concurrent any other cancer (except BCC or squamous cell carcinoma of skin).
2. Inability to adhere to monthly visits to the oncology unit for evaluation.
3. Presence of brain metastases.
4. Any current or recent (within the last month) continuous treatment by steroids or by NSAIDs, or with therapeutic doses of anticoagulants for any reason.
5. Previous radiotherapy to the only site of measurable disease.
6. Evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac including arrhythmias, hepatic or renal disease), and/or existence of active peptic ulcer (clinically and/or by gastroscopy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Length of progression free survival (PFS), measured in months. | Up to 12 months.
  From start of the experimental treatment until the date of first documented progression or date of death of any cause,whichever came first, assessed up to 12 months.

SECONDARY OUTCOMES:
Toxicity profile of treatment, defined by CTCAE Version 4.0. | up to12 months
  From start of the experimental treatment until the date of first documented progression or date of death of any cause,whichever came first, assessed up to 12 months.
Changes in levels of angiogenic factors while under treatment: VEGF, PDGF, TSP-1 | Up to 4 months.
  Change from baseline in levels of angiogenic factors at 4 months of treatment.
Quality of life, as expressed by FACT-C. | Up to 12 months.
  Change from baseline in parameters of Quality of life until the end of treatment, assessed up to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: David Loven, MD, Principal Investigator — Ha'Emek MC
Locations (1):
- HaEmek Medical Center, Afula, Israel